CLINICAL TRIAL: NCT05538325
Title: After the End of the Puerperium: Kinematic Assessment of Lumbar Spine Active Range of Motion in Women Who Experienced Cesarean or Vaginal Birth
Brief Title: Assessment of Lumbar Spine Active Range of Motion in Women Who Were Experienced Cesarean or Vaginal Birth
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Abouelyazeed Ali, Lecturer of Physical Therapy for Women's Health, South Valley University
Other Study IDs: Lumbar Spine ROM
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-09

CONDITIONS: Cesarean and Vaginal Birth Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group A: 25 females who experienced cesarean birth
  Interventions: Device: Bubble Inclinometer and Digital Pelvic Inclinometer
- Group B: 16 females who experienced vaginal birth
  Interventions: Device: Bubble Inclinometer and Digital Pelvic Inclinometer
- Group C: 25 females who were the controls, did not experience any pregnancy
  Interventions: Device: Bubble Inclinometer and Digital Pelvic Inclinometer

INTERVENTIONS:
Device: Bubble Inclinometer and Digital Pelvic Inclinometer — They are valid and reliable devices to measure the range of motion of the lumbar spine

SUMMARY:
Pregnancy may impact the musculoskeletal apparatus of females through pregnancy-associated biomechanical, vascular, and hormonal changes. Pregnant females may complain of lumbopelvic pain, especially during their last trimester. This lumbopelvic pain can be the result of an enlarged uterus and unstable lumbopelvic joints.

DETAILED DESCRIPTION:
Cesarean birth can affect the lumbopelvic biomechanics through its impact on the sacroiliac joints and the abdominal muscles. while vaginal birth can trigger lumbopelvic pain through its impact on the pelvic joints like the symphysis pubis and sacroiliacs.

When puerperium is finished, most of these pregnancy-related changes assume its prepregnant conditions.

Physiotherapists are responsible for providing PT care for women to improve their quality of life during the puerperium and even during the delayed postpartum interval.

ELIGIBILITY:
Inclusion Criteria:

1. All women either primiparous or multiparous have not had anaesthesia (epidural, spinal, or general) for at least one year prior to the last obstetric anaesthesia.
2. Their ages ranged from 18 to 35 years.
3. Participants were assessed between the 6th week to the 12th week postnatal.
4. All participants were able to continue all assessment procedures.
5. They might have a mild or moderate myofascial LBP

Exclusion Criteria:

1. Women who were below 18 years old or above 35 years.
2. Women who did not continue all assessment procedures.
3. Women who had a severe myofascial LBP or any specific low back conditions.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — It is a study for investigation of cesarean or vaginal birth complications on the lumbar spine movements after the end of puerperium
Study Population: 66 women participated in this study. They were recruited from the Woman and Child Hospital of South Valley University, located in Qena governorate, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
Lumbar Spine Extension Active Range of Motion | Assessment will be done 6-12 weeks after Cesarean or Vaginal birth
  It represent the non-painful full range of motion from standing upright to leaning backward in the sagittal plane
Lumbar Spine Flexion Active Range of Motion | Assessment will be done 6-12 weeks after Cesarean or Vaginal birth
  It represent the non-painful full range of motion from standing upright to leaning forward in the sagittal plane
Lumbar Spine Right Side Bending Active Range of Motion | Assessment will be done 6-12 weeks after Cesarean or Vaginal birth
  It represent the non-painful full range of motion from standing upright to leaning sideway to the right in the frontal plane
Lumbar Spine Left Side Bending Active Range of Motion | Assessment will be done 6-12 weeks after Cesarean or Vaginal birth
  It represent the non-painful full range of motion from standing upright to leaning sideway to the left in the frontal plane
Lumbar Spine Right Axial Rotation Active Range of Motion | Assessment will be done 6-12 weeks after Cesarean or Vaginal birth
  It represents the non-painful full range of motion from standing with trunk forward bended 90 degree then head, neck, shoulders, and trunk rotation to the right side
Lumbar Spine Left Axial Rotation Active Range of Motion | Assessment will be done 6-12 weeks after Cesarean or Vaginal birth
  It represents the non-painful full range of motion from standing with trunk forward bended 90 degree then head, neck, shoulders, and trunk rotation to the left side

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, South Valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thabah M, Ravindran V. Musculoskeletal problems in pregnancy. Rheumatol Int. 2015 Apr;35(4):581-7. doi: 10.1007/s00296-014-3135-7. Epub 2014 Sep 25. PMID 25253297
- [Background] Kesikburun S, Guzelkucuk U, Fidan U, Demir Y, Ergun A, Tan AK. Musculoskeletal pain and symptoms in pregnancy: a descriptive study. Ther Adv Musculoskelet Dis. 2018 Nov 19;10(12):229-234. doi: 10.1177/1759720X18812449. eCollection 2018 Dec. PMID 30515249
- [Background] Ritchie JR. Orthopedic considerations during pregnancy. Clin Obstet Gynecol. 2003 Jun;46(2):456-66. doi: 10.1097/00003081-200306000-00024. No abstract available. PMID 12808395
- [Background] Franklin ME, Conner-Kerr T. An analysis of posture and back pain in the first and third trimesters of pregnancy. J Orthop Sports Phys Ther. 1998 Sep;28(3):133-8. doi: 10.2519/jospt.1998.28.3.133. PMID 9742469
- [Background] Sung S, Mahdy H. Cesarean section. InStatPearls [Internet] 2021 Apr 25. StatPearls Publishing.
- [Background] Sanya AO, Olajitan A. Comparison of abdominal muscle strength in post-parous and nil parous subjects. Afr J Med Med Sci. 1999 Mar-Jun;28(1-2):49-53. PMID 12953987
- [Background] Fan C, Guidolin D, Ragazzo S, Fede C, Pirri C, Gaudreault N, Porzionato A, Macchi V, De Caro R, Stecco C. Effects of Cesarean Section and Vaginal Delivery on Abdominal Muscles and Fasciae. Medicina (Kaunas). 2020 May 27;56(6):260. doi: 10.3390/medicina56060260. PMID 32471194
- [Background] Ghodke PS, Shete D, Anap D. Prevalence of sacroiliac joint dysfunction in postpartum women-a cross sectional study. Physiother Rehabil. 2017;2(3):149.